CLINICAL TRIAL: NCT02576587
Title: Elucidation of the Influence of Sleep Apnea on Risk of Atrial Fibrillation
Brief Title: Influence of Sleep Apnea on Risk of Atrial Fibrillation
Acronym: Safebeat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Reena Mehra, MD, Director of Sleep Disorders Reseach, Associate Professor of Medicine, The Cleveland Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-594; R01HL109493 (NIH)
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Sleep Apnea; Atrial Fibrillation
MeSH Terms: conditions — Sleep Apnea Syndromes; Atrial Fibrillation | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case (diagnosed with PAF) (Other): Cases. Patients with Paroxysmal Atrial Fibrillation who present to Electrophysiology Clinic at UHCMC and the Cleveland Clinic Foundation will be approached for recruitment in the study.
  Cases found to have an apnea hypopnea index >=15 will be asked to continue in the study for 3 months wearing a Continuous Positive Airway Pressure (CPAP) machine.
  Interventions: Other: Continuous Positive Airway Pressure
- Controls (No Intervention): Controls. Patients without AF will be recruited from General Cardiology and Internal Medicine clinics (geographically similar to controls). Selection bias will be minimized as there are a broad range of reasons for patients to present to these clinics.

INTERVENTIONS:
Other: Continuous Positive Airway Pressure — For cases, those found to have moderate sleep apnea (AHI >=15) will be place on CPAP therapy.
  Arms: Case (diagnosed with PAF)

SUMMARY:
The Elucidation of the Influence of Sleep Apnea on Risk of Atrial Fibrillation study.

The study involves a case control design to investigate the extent to which there is an independent relationship of sleep disordered breathing (SDB) and paroxysmal atrial fibrillation (PAF). Cases will be defined as clinically identified patients with PAF and controls as those without AF. In order to rigorously address important biologic confounding influences, the cases and controls will be individually matched based upon age, gender, race, and body mass index. Those participants with both PAF and SDB (Apnea Hypopnea Index, AHI>=15) will be asked to return for a follow up exam after 3 months of SDB treatment in the Clinical Research Unit (CRU) for collection of the same measures collected at the baseline exam to observe for any significant changes with the purpose of collecting effect size data to inform future clinical trials.

The total duration of the study is 4 years. The duration for any individual participant is up to from one to 13 weeks months, including a 3-month treatment period for those with moderate to severe SDB, i.e. AHI>15.

DETAILED DESCRIPTION:
Sleep-disordered breathing (SDB) is common in patients with cardiovascular disease and its attendant hypoxemia and autonomic dysfunction create a milieu that is likely to enhance AF propensity. Thus, SDB may represent a novel target for AF prevention and treatment strategies. Although our prior cross-sectional work has shown a 2-4 fold higher odds of AF related to SDB, these and other reports have not included cardiac structural data or autonomic/biochemical measures, and have addressed only arrhythmic events occurring during an overnight sleep study. In this proposal, we will examine paroxysmal AF (PAF), an early stage risk factor for persistent AF, and relevant to this proposal because it occurs prior to extensive cardiac electrical remodeling/fibrosis.

OUTLINE OF STUDY VISITS Baseline Visit (SA 1 and 2). After informed consent, eligible participants will be scheduled to arrive for an overnight visit in the CRU. During the evening, participants will undergo questionnaire administration, blood pressure measurements, and anthropometry. They will be provided dinner and undergo polysomnography (PSG). In the morning, participants will undergo fasting venipuncture, overnight urine collection, ECHO, 6 minute walk test, vascular measures and blood pressure measurements. For those with PAF (cases), hook-up for continuous ECG monitoring will be performed along with education regarding how to handle the device and bathing instructions, etc. All measurements in the DCRU/CRU will be performed blinded to PAF status. The only unblinded staff will be a dedicated research assistant who will perform the ECG monitoring hook-up. Blinded staff will collect and process data and perform data entry. After the baseline visit, participants with PAF (n=150) will undergo hook-up of the ECG monitor and an activity monitor at the baseline visit to wear for a 7-21 day period.

Follow-Up Visit (SA3). Those with SDB (AHI>=15) without evidence of central apnea (central apnea index>5) or Cheyne Stokes Respirations via baseline visit PSG and who have PAF will undergo the following. A 5-7 day home-based auto-titration (APAP, Respironics Autopap System One with humidifier) to identify the optimal positive airway pressure (PAP) setting will be performed (with settings 4-20cm H2O). At the end of the 5-7 day titration, the goal will be to identify the pressure that results in an AHI<5 events/hour (optimally). The research assistant will re-set the device to deliver this optimal fixed pressure identified by the PI through the secure wireless web-site. An overnight DCRUCRU visit will be scheduled after 3 months of wearing CPAP during which the same measures performed at the baseline visit will be collected.

STUDY PROCEDURES 2-DIMENSIONAL DOPPLER ECHOCARDIOGRAPHY. Parasternal, apical and subcostal 2-D views and apical 3D views will be obtained with transducer orientation and gain settings adjusted to optimally define endocardial surface of each cardiac chamber.

POLYSOMNOGRAPHY (PSG). Procedure for PSG: Research PSG will be performed using the Compumedics E-series system (Abbottsford, AU) which will include 3 cortical encephalograms, bilateral electro-oculograms, a bipolar submental electromyogram, thoracic and abdominal respiratory inductance plethysmography, airflow (by nasal-oral thermocouple and nasal cannula pressure recording), oximetry (using highly sensitive finger pulse oximeter, sampling frequency 25Hz), electrocardiogram (ECG) at 250Hz (used to derive HRV measures of autonomic function); body position (mercury switch sensor), bilateral leg movements. EEGs are recorded at 125Hz. 3) 7-21 Day CONTINUOUS ECG MONITORING.

Procedure: A 3-lead (2 channel), wireless, lightweight ECG monitoring device will be used to collect the ECG data over a 7-21 day period in those with PAF after the baseline and follow-up CRU visits.

ACTIVITY MONITORING. Procedure: An accelerometer (GT3X+, Actigraph Co., Ft Walton Bch, Fl) will be used for 7-21 days, coincident with the time of continuous ECG monitoring.

FASTING VENIPUNCTURE (52cc). Procedure: Phlebotomy will be performed the morning of the baseline and follow-up visits using standard techniques by trained research staff following written procedures. 6) DNA collection. Blood will be collected to extract RNA, which will be stored to test future hypotheses regarding genetic determinants of treatment response.

OVERNIGHT URINE. Procedure: Overnight urine collection will be performed. ANTHROPOMETRY. Height (inches, cm), neck circumference (cm), waist circumference (cm), hip circumference (cm) will be obtained. Skinfolds are measured with calibrated metal calipers from 7 sites (chest, calf, thigh, calf, subscapular, midaxillary, suprailiac, abdominal).

RESTING BLOOD PRESSURE (BP). BP will be measured after the participant has been sitting quietly for at least 5 minutes following standardized guidelines using a calibrated sphygmomanometer. Measurements will be repeated three times and recorded.

QUESTIONNAIRES. The following will be collected: a) The Berlin Sleep Questionnaire, b) Epworth Sleepiness Scale, c) The Sleep Habits and Medical Condition Questionnaire d) The Medical Outcomes Survey-SF 36 (MOS-SF) e) Patient Health Questionnaire-9 (PHQ-9) f) Daily ECG/Activity Log g) Atrial Fibrillation Effect on Quality-of-life, a 20-item questionnaire that assesses the impact of atrial fibrillation on quality of life.

6 Minute Walk Test. Baseline oxygen saturation and heart rate will be recorded. If oxygen saturation >90%, then proceed with protocol. Using the BORG Scale record rate the symptoms of breathlessness and leg fatigue after a 6 minute walk at usual pace.

Arterial Applanation Tonometry: Radial artery measurements will be performed after sphygmomanometric pressure is obtained with use of an applanation tonometry probe with a minimum of two consecutive measurements to obtain pulse wave analysis results. For pulse wave velocity, lead II ECG will be performed along with cardotid and femoral applanation tomometry.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Cases:

PAF defined by recurrent episodes of AF, which self-terminate within a 7-day period (based upon AHA consensus statement 77)

Age 18-80 years

Individuals able to participate in > 2 overnight/daytime sleep and physiologic assessments over a 3 month period.

Inclusion Criteria for Controls:

Age 18 to 80 years

Individuals in normal sinus rhythm (NSR) with no current AF or history of AF

Individuals able to participate in an overnight/daytime sleep and physiologic assessment.

Exclusion Criteria:

Exclusion Criteria for Cases:

PAF with rapid or uncontrolled rate (>120bpm)

Post-operative PAF

History of cardiac ablation or successful electro-cardioversion for PAF (ablation for other arrhythmias such as AVNRT and if PAF persists after cardioversion is acceptable )

Valvular stenosis, prosthesis or significant valvular insufficiency [i.e. those with moderate or greater severity of aortic stenosis (aortic valve area <1.5 cm2), mitral regurgitation which is moderate or more severe in degree (>20% regurgitant fraction) or moderate or greater severity mitral stenosis (mitral valve area <1.5 cm2)]

Atrial septal defect

Infiltrative/restrictive cardiomyopathy

Sick sinus syndrome

Previously diagnosed SDB on specific SDB treatments (CPAP, oral appliances)

Severe chronic insomnia

Circadian rhythm disorder (e.g. shift work sleep disorder, delayed or advanced sleep phase syndrome)

Insufficient sleep syndrome defined by reported sleep duration < 4 hrs

Supplemental oxygen use

Unstable medical conditions (e.g., new onset or changing angina, a myocardial infarction or congestive heart failure exacerbation documented within the previous 3 months, systolic heart failure (Left Ventricular Ejection Fraction < 35%), high grade cardiac dysrhythmia/heart block, stroke with functional limitations, uncontrolled hypertension (BP>170/110), abdominal aneurysm >5.5 cm or >1 cm growth/year, uncontrolled diabetes mellitus (HbA1c>9.0), pulmonary hypertension, non-skin cancer diagnosis or treatment within the previous year, end stage renal and hepatic failure, immunodeficiencies (HIV, HCV), uncontrolled hypo- or hyperthyroidism)

Psychiatric disorders which are inadequately treated

Compromised competence

Alcohol abuse (currently drinks >5 alcoholic drinks/day)

Pregnancy

Inability to provide informed consent

Illicit drug use over last 6 months

Rate controlling anti-arrhythmic medication (Classes I-III and V) with no further clinical occurrence of PAF

Has a Pacemaker or Implantable cardioverter-defibrillator.

Rationale for criteria: The goal of this study is to include those patients with PAF that is not secondary to the post-operative period or valvular disease and without ablation as these processes would result in alteration of atrial physiology and preclude assessment of independent SDB effects on AF which is independent of these conditions. Patients with sleep disorders will be excluded as sleep disorders may influence arrhythmogenesis. Those on treatment for SDB will be excluded because treatment would preclude assessment of SDB pathophysiologic effects on atrial arrhythmogenesis. Those with unstable medical conditions or rapid or uncontrolled heart rate will be excluded due to safety reasons.

Note: Exclusion criteria for positive airway pressure (PAP) intervention: Central Apnea Index>5 noted on baseline examination sleep study or evidence of Cheyne Stokes Respirations/periodic breathing (cyclical crescendo and decrescendo change in breathing amplitude).

Exclusion Criteria for Controls:

Current or history of AF, otherwise the same exclusion criteria listed for cases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reena Mehra, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] May AM, Wang L, Kwon DH, Van Wagoner DR, Chung MK, Dalton JE, Mehra R. Sleep apnea screening instrument evaluation and novel model development and validation in the paroxysmal atrial fibrillation population. Int J Cardiol Heart Vasc. 2020 Sep 4;31:100624. doi: 10.1016/j.ijcha.2020.100624. eCollection 2020 Dec. PMID 33364332

RESULTS

PARTICIPANT FLOW:
Groups:
- Case (Diagnosed With PAF): Cases. Patients with Paroxysmal Atrial Fibrillation who present to Electrophysiology Clinic at UHCMC and the Cleveland Clinic Foundation will be approached for recruitment in the study.
  Cases found to have an apnea hypopnea index >=15 will be asked to continue in the study for 3 months wearing a Continuous Positive Airway Pressure (CPAP) machine.
  Continuous Positive Airway Pressure: For cases, those found to have moderate sleep apnea (AHI >=15) will be place on CPAP therapy.
Period: Baseline
Arm/Group | Case (Diagnosed With PAF) | Controls
Started | 161 (Total cases baseline visit) | 156 (Total controls baseline visit)
Completed | 161 (Baseline visit completed) | 155 (Baseline visit completed)
Not Completed | 0 | 1
Not completed — Equipment failure | 0 | 1
Period: Follow up Period (Case Only)
Arm/Group | Case (Diagnosed With PAF) | Controls
Started | 161 (Completed baseline.) | 155 (Controls not eligible for follow-up)
Selected for Follow up (Cases with apnea hypopnea index greater or equal to 15 were selected for follow up.) | 61 | 0
Completed | 44 | 0
Not Completed | 117 | 155
Not completed — Withdrawal by Subject | 25 | 0
Not completed — Not selected for follow up (AHI<15) | 92 | 0
Not completed — Controls not eligible for followup | 0 | 155

BASELINE CHARACTERISTICS:
Population: Cases and controls completed baseline visit and having matched controls/cases were included in baseline analysis.
Groups:
- Case (Diagnosed With PAF): Cases. Patients with Paroxysmal Atrial Fibrillation who present to Electrophysiology Clinic at UHCMC and the Cleveland Clinic Foundation will be approached for recruitment in the study.
  Cases completed baseline and having matched controls were included in baseline data analysis.
- Controls: Controls. Patients without AF will be recruited from General Cardiology and Internal Medicine clinics (geographically similar to controls). Selection bias will be minimized as there are a broad range of reasons for patients to present to these clinics.
  Controls completed baseline and having matched cases were included in baseline data analysis.
- Total: Total of all reporting groups
Arm/Group | Case (Diagnosed With PAF) | Controls | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12) | 62 (12) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 95 | 95 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 149 | 149 | 298
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 22 | 44
  White | 125 | 125 | 250
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31 (7) | 32 (7) | 31 (7)
Apnea Hypopnea Index (AHI) [Median (Inter-Quartile Range); unit: apneas plus hypopneas per hour] — AHI equals number of apnea and hypopnea breathing pauses divided by sleep duration in hours. It has a lower limit zero, but no upper limit. Greater AHI indicates higher severity of sleep apnea. The AHI values for adults are categorized as:
  Normal: AHI<5; Mild sleep apnea: AHI greater than or equal to 5 and <15; Moderate sleep apnea: AHI greater than or equal to 15 and <30; Severe sleep apnea: any AHI value greater than or equal to 30.
  In this study, cases having AHI greater than or equal to 15 qualifies for follow-up.
  apneas plus hypopneas per hour | 11 [4 to 24] | 13 [4 to 24] | 12 [4 to 24]
Arousal Index [Median (Inter-Quartile Range); unit: Arousals per hour] — Arousal index (AI) equals number of arousals divided by sleep duration in hours. Arousals are interruptions of sleep lasting 3 to 15 seconds, spontaneously or as a result of sleep disordered breathing or other sleep disorders. It has a lower limit zero, but no upper limit. The range of AI for adults varies by age, e.g. 10-12/hour are normal at age 20, 20-22/hour are normal at age 50-60.
  Arousals per hour | 18 [13 to 26] | 19 [13 to 28] | 19 [13 to 27]
Central Apnea Index [Median (Inter-Quartile Range); unit: Central apneas per hour] — Central apnea index (CAI) equals number of central apneas divided by sleep duration in hours. Greater central apnea index indicates higher severity of sleep apnea. It has a lower limit zero, but no upper limit. The CAI values for adults are categorized as:
  Normal: CAI<5; Mild sleep apnea: CAI greater than or equal to 5 and <15; Moderate sleep apnea: CAI greater than or equal to 15 and <30; Severe sleep apnea: any CAI value greater than or equal to 30.
  Central apneas per hour | 0 [0 to 0.4] | 0 [0 to 0.4] | 0 [0 to 0.4]
Percent sleep time with oxygen saturation<90% [Median (Inter-Quartile Range); unit: percent of sleep time] | 0.4 [0 to 3] | 0.4 [0 to 2] | 0.4 [0 to 3]
Left Atrial Volume [Median (Inter-Quartile Range); unit: mL] — Increased left atrial volume and strain are known risk factors of AF and PAF. Population: Echocardiography measurements were not available for some subjects due to image quality. If at least one of the matched case and control had missing value, this pair of subjects was not included in analysis.
  mL
    number analyzed (Participants) | 135 | 135 | 270
    (all) | 63 [48 to 77] | 51 [45 to 71] | 60 [46 to 75]
Left Atrial Volume Index [Median (Inter-Quartile Range); unit: mL/m^2] — Increased left atrial volume and strain are known risk factors of AF and PAF. Left atrial volume index (LAVI) is left atrial size indexed to Body surface area (BSA). The reference range of LAVI is 16-28 mL/m^2.
  Mildly abnormal: 29-33 mL/m^2; Moderately abnormal: 34-39 mL/m^2; Severely abnormal: greater than or equal to 40 mL/m^2. Population: Echocardiography measurements were not available for some subjects due to image quality. If at least one of the matched case and control had missing value, this pair of subjects was not included in analysis.
  mL/m^2
    number analyzed (Participants) | 134 | 134 | 268
    (all) | 30 [23 to 37] | 28 [22 to 33] | 29 [23 to 35]
Left Atrial Systolic Strain by apical four-chamber (A4C) view [Median (Inter-Quartile Range); unit: percent of left atrial volume] — Left atrial systolic strain, a measure of left atrial remodeling which is inversely related to fibrosis in PAF, is measured by 2-dimensional echocardiography. Apical four-chamber and two-chamber views are the most commonly used approaches to measure the strain rate (%) of left atrial. Population: Echocardiography measurements were not available for some subjects due to image quality. If at least one of the matched case and control had missing value, this pair of subjects was not included in analysis.
  percent of left atrial volume
    number analyzed (Participants) | 107 | 107 | 214
    (all) | 34 [25 to 40] | 33 [27 to 41] | 33 [27 to 41]
Left Atrial Systolic Strain by apical two-chamber (A2C) view [Median (Inter-Quartile Range); unit: percent of left atrial volume] — Left atrial systolic strain, a measure of left atrial remodeling which is inversely related to fibrosis in PAF, is measured by 2-dimensional echocardiography. Apical four-chamber and two-chamber views are the most commonly used approaches to measure the strain rate (%) of left atrial. Population: Echo measurements were not available for some subjects due to image quality. If at least one of the matched case and control had missing value, this pair of subjects was not included in analysis.
  percent of left atrial volume
    number analyzed (Participants) | 106 | 106 | 212
    (all) | 34 [29 to 41] | 35 [29 to 43] | 35 [29 to 42]
High Blood Pressure or Hypertension [Count of Participants; unit: Participants] | 87 | 79 | 166
High Blood cholesterol [Count of Participants; unit: Participants] | 86 | 91 | 177
History of heart attack [Count of Participants; unit: Participants] | 9 | 16 | 25
Depression [Count of Participants; unit: Participants] | 22 | 35 | 57
Diabetes [Count of Participants; unit: Participants] | 19 | 23 | 42
Use of Calcium blocker [Count of Participants; unit: Participants] | 20 | 8 | 28
Use of beta blocker [Count of Participants; unit: Participants] | 85 | 35 | 120
Any use of antihypertension medications [Count of Participants; unit: Participants] — Medications included Ace Inhibitors, Antihypertensive, Alpha-2 Blocker, Beta-Blocker, Calcium blocker, Diuretic and Nitrates.
  Participants | 121 | 69 | 190

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Paroxymal Atrial Fibrillation (PAF)
Description: Patients with diagnosis of PAF were defined as cases. PAF is the primary outcome of baseline analysis, which aimed to quantify the association of sleep apnea and PAF.
Time Frame: Baseline
Population: Cases and controls who had matched control/case were included in baseline analysis. Only 150 cases were one-to-one matched with controls.
Measure: Count of Participants; unit: Participants
Arm/Group | Case (Diagnosed With PAF) | Controls
Number analyzed (Participants) | 150 | 150
Participants | 150 | 0
Statistical Analysis 1: Comparison: Case (Diagnosed With PAF) vs Controls; Test type: Other — Conditional logistic regression was used to assess the relationship of PAF and AHI on matched pairs of case and control; p = 0.054, Conditional logistic regression; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.97 to 1.00], Standard Error of Mean 0.007
Statistical Analysis 2: Comparison: Case (Diagnosed With PAF) vs Controls; Test type: Other — Conditional logistic regression was used to assess the relationship of PAF and LA volume on matched pairs of case and control; p = 0.014, Conditional logistic regression; N = 270 (135 cases and 135 controls); Odds Ratio (OR) = 1.02, 95% CI 2-sided [1.00 to 1.03], Standard Error of Mean 0.007
Statistical Analysis 3: Comparison: Case (Diagnosed With PAF) vs Controls; Test type: Other — Conditional logistic regression was used to assess the relationship of PAF and LA volume index on matched pairs of case and control; p = 0.030, Conditional logistic regression; N=268 (134 cases and 134 controls); Odds Ratio (OR) = 1.03, 95% CI 2-sided [1.00 to 1.06], Standard Error of Mean 0.015
Statistical Analysis 4: Comparison: Case (Diagnosed With PAF) vs Controls; Test type: Other — Conditional logistic regression was used to assess the relationship of PAF and LA systolic strain apical four-chamber (A4C) on matched pairs of case and control; p = 0.39, Conditional logistic regression; N=214 (107 cases and 107 controls); Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.96 to 1.01], Standard Error of Mean 0.013
Statistical Analysis 5: Comparison: Case (Diagnosed With PAF) vs Controls; Test type: Other — Conditional logistic regression was used to assess the relationship of PAF and LA systolic strain apical two-chamber (A2C) on matched pairs of case and control; p = 0.49, Conditional logistic regression; N=212 (106 cases and 106 controls); Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.97 to 1.02], Standard Error of Mean 0.013

2. Secondary Outcome: Echocardiography Measures- Left Atrial Volume
Description: Increased left atrial volume and strain are known risk factors of AF and PAF. Echocardiography measurements were not available for some subjects due to image quality.
Time Frame: Baseline and 12 week follow up
Population: Cases found to have an apnea hypopnea index >=15 were asked to continue in the study for 3 months wearing a Continuous Positive Airway Pressure (CPAP) machine.
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Case Baseline: Case baseline measurements
- Case Follow-up: Case follow-up measurements
Arm/Group | Case Baseline | Case Follow-up
Number analyzed (Participants) | 43 | 39
mL | 67 [52 to 79] | 72 [55 to 80]
Statistical Analysis 1: Comparison: Case Baseline vs Case Follow-up; Test type: Other; p = 0.16, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test was used to compare pre- and post- treatment outcomes; median of change = 3.4; Inter-Quartile Range of the change (post minus pre) is (-7.0, 13.7)

3. Secondary Outcome: Echocardiographic Measures- LA Volume Index
Description: Increased left atrial volume and strain are known risk factors of AF and PAF. Left atrial volume index (LAVI) is left atrial size indexed to Body surface area (BSA). The reference range of LAVI is 16-28 mL/m^2.
  Mildly abnormal: 29-33 mL/m^2; Moderately abnormal: 34-39 mL/m^2; Severely abnormal: greater than or equal to 40 mL/m^2.
  Echocardiography measurements were not available for some subjects due to image quality.
Time Frame: Baseline and 12 week follow up
Measure: Median (Inter-Quartile Range); unit: mL/m^2
Arm/Group | Case Baseline | Case Follow-up
Number analyzed (Participants) | 42 | 38
mL/m^2 | 31 [23 to 37] | 30 [24 to 38]
Statistical Analysis 1: Comparison: Case Baseline vs Case Follow-up; Test type: Other; p = 0.088, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test was used to compare pre- and post- treatment outcomes; median of change = 1.8 — Inter-quartile range of the change (post minus pre) is (-2.0, 6.0)

4. Secondary Outcome: Echocardiographic Measures- LA Systolic Strain by A4C View
Description: Left atrial systolic strain, a measure of left atrial remodeling which is inversely related to fibrosis in PAF, is measured by 2-dimensional echocardiography. Apical four-chamber (A4C) and two-chamber (A2C) views are the most commonly used approaches to measure the strain rate (%) of left atrial.
Time Frame: Baseline and 12 week follow up
Measure: Median (Inter-Quartile Range); unit: percentage of left atrial volume
Arm/Group | Case Baseline | Case Follow-up
Number analyzed (Participants) | 34 | 32
percentage of left atrial volume | 36 [24 to 46] | 29 [23 to 38]
Statistical Analysis 1: Comparison: Case Baseline vs Case Follow-up; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test was used to compare pre- and post- treatment outcomes; median of change = -3.7 — Inter-quartile range of the change (post minus pre) is (-8.0, -0.57)

5. Secondary Outcome: Echocardiographic Measures- LA Systolic Strain by A2C View
Description: as for outcome 4
Time Frame: Baseline and 12 week follow up
Measure: Median (Inter-Quartile Range); unit: percentage of left atrial volume
Arm/Group | Case Baseline | Case Follow-up
Number analyzed (Participants) | 34 | 31
percentage of left atrial volume | 36 [27 to 41] | 37 [28 to 45]
Statistical Analysis 1: Comparison: Case Baseline vs Case Follow-up; Test type: Other; p = 0.59, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test was used to compare pre- and post- treatment outcomes; median of change = -0.70 — Inter-quartile range of the change (post minus pre) is (-6.2, 10.7)

6. Secondary Outcome: Vascular Measures- Pulse Wave Velocity
Description: Radial measurements were performed on the same arm using the SphygmoCor device after sphygmomanometric pressure was obtained with use of an applanation tonometry probe containing a solid state high fidelity Millar transducer over the radial artery with a minimum of two consecutive measurements to obtain pulse wave analysis results. For pulse wave velocity, lead II ECG (LL, LA, RA) was performed along with cardotid and femoral applanation tomometry. Orientation and pressure applied to the transducer were adjusted to optimize applanation of the artery between the transducer and the underlying tissue. Waveforms were processed using the SphygmoCor software (model EM3, version CvMS 9.0, Atcor Medical Pty, West Ryde, Australia).)
Time Frame: Baseline and 12 week follow up
Population: Cases selected for follow-up and having available SphygmoCor measurements
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Case Baseline | Case Follow-up
Number analyzed (Participants) | 14 | 10
m/s | 9.5 (2.7) | 10.5 (3.8)
Statistical Analysis 1: Comparison: Case Baseline vs Case Follow-up; Test type: Other; p = 0.65, t-test, 2 sided; Paired t test was used to compare pre- and post- treatment outcomes; mean of change = 0.62, Standard Deviation 4.2

7. Secondary Outcome: Vascular Measures- Augmentation Index
Description: Augmentation Index (Alx) is an indication of systemic arterial stiffness and measures the contributions of wave reflection to central systolic pressure. Scores vary based on age and gender and in a normal, healthy population research has shown can range from -10% or less up to 50%. A negative augmentation index suggests low artery stiffness (late arriving wave reflections) and a positive index is a reflection of increase artery stiffness (reflective wave arriving early in the cardiac cycle). Waveforms will be processed using the SphygmoCor software (model EM3, version CvMS 9.0, Atcor Medical Pty, West Ryde, Australia) for this measurement.
  It is calculated at the onset of reflected wave, Alx = AP/PP x 100. Alx = Augmentation Index, the percentage of the pulse pressure due to the AP; PP = Pulse Pressure; AP = Augmentation Pressure, the contribution of the reflected wave to the pulse pressure.
Time Frame: Baseline and 12 week follow up
Population: Cases selected for follow-up and having available SphygmoCor measurements
Measure: Mean (Standard Deviation); unit: percentage of augmentation pressure
Arm/Group | Case Baseline | Case Follow-up
Number analyzed (Participants) | 17 | 17
percentage of augmentation pressure | 28.6 (13.2) | 26.9 (11.6)
Statistical Analysis 1: Comparison: Case Baseline vs Case Follow-up; Test type: Other; p = 0.65, t-test, 2 sided; Paired t test was used to compare pre- and post- treatment outcomes; mean of change = -1.7, Standard Deviation 12.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all participants during their overnight visit. Participants (cases) which qualified for CPAP, adverse events were collected over a 3 month period while wearing CPAP.
Arm/Group | Case (Diagnosed With PAF) | Controls
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/155
Serious Adverse Events (participants affected / at risk) | 7/161 | 0/155
Other Adverse Events (participants affected / at risk) | 22/161 | 0/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Case (Diagnosed With PAF) (N=161) | Controls (N=155)
Hit by Automobile (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — visit to ER
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Headache from prior car accident
Elective Tummy Tuck Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective Ablation for Atrial Fibrillation (Surgical and medical procedures) | 1 (1) | 0 (0)
High Blood Pressure (went to ER) (Cardiac disorders) | 1 (1) | 0 (0)
Obstructed Bowel (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalized
Elective - Total Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Case (Diagnosed With PAF) (N=161) | Controls (N=155)
Muscle and skeletal pain from Echocardiogram (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Itching/inflammation fron ECG pads (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) — (From wearing continuous ECG)
Itching head from CPAP headwear (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Poison Ivy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Heart Rate 130-190 bpm (Cardiac disorders) | 1 (1) | 0 (0) — (Alerted form continuous ECG Monitor) Forgot to take medication.
Injured Knee in shower (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nail puctured hand (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Runny nose with CPAP use (General disorders) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Bloody nose (slight) upon wakening (General disorders) | 1 (1) | 0 (0) — (with CPAP use)
Twisted ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Continuous ECG Alert (Cardiac disorders) | 1 (1) | 0 (0) — (A-fib noted)
A-Fib went to ER (Cardiac disorders) | 1 (1) | 0 (0)
Fell off motorcycle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — cracked rib
A-fib with shortness of breath (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT02576587/Prot_SAP_000.pdf